# Are Sugar-Sweetened Beverage Information Labels Well-Targeted? NCT05038163

Study Protocol August 17<sup>th</sup>, 2021

#### Protocol # 2020-08-13558 Date Printed: 08/17/2021

| Personnel Information | 1 |
|-----------------------------------------|----|
| Vulnerable Subject Checklist | 3 |
| Study Sites | 4 |
| General Checklist | 5 |
| Funding | 6 |
| Exempt Paragraph(s) | 8 |
| Purpose,Study Procedures and Background | 12 |
| Subject Population | 19 |
| Risks | 20 |
| Procedures to Maintain Confidentiality | 22 |
| Attachments | 24 |
| Assurance | 26 |
| Event History | 28 |

Protocol # 2020-08-13558 Date Printed: 08/17/2021

Protocol Title:

Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened

beverages

Protocol Type:

Soc-Behav-Ed Exempt

Date Submitted:

06/27/2021

Important Note:

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

### \* \* \* Personnel Information \* \* \*

Enter all study personnel (if not previously entered) and relevant training information. Please read Personnel Titles and Responsibilities: Roles in eProtocol before completing this section.

Note: The Principal Investigator or Faculty Sponsor, Co-Principal Investigator, Student or Postdoctoral Investigator, Administrative Contact, and Other Contact can EDIT and SUBMIT. Other Personnel can only VIEW the protocol.

Principal Investigator or Faculty

**Email** 

Name of Principal Investigator

Degree (e.g., MS/PhD)

Title Dr

Fax

Dmitry Taubinsky

Phone

dmitry.taubinsky@berkeley.edu

7074808125

Department Name

Malling Address

**Economics** 

94720

UCB status (select all that apply):

X Faculty Postdoc

Grad

Undergrad Other

Faculty (with some exceptions), staff, and students engaged in human subjects research must complete either the biomedical or social-behavioral human research course through the online Collaborative Institutional Training Initiative (CITI), depending upon which is most germane to the research. ALL PIs on an NIH award are required to complete either CITI or NIH Training. See Training and Education for more information.

If applicable, please insert date (mm/dd/vv) of completion in appropriate box(es) below:

| ii applicable, picase ilisei | t date (minadayy) of completion in appr | ophate box(es) below. |
|---|---|---|
| CITI | NIH | Other Training (title & date completed) |
| 12/29/17 | | |

#### Student or Postdoctoral Investigator

NOTE: All Student/Postdoc Investigators must have a Faculty Sponsor who will serve as the "responsible researcher." If NOT a student or postdoc project, enter student(s) and/postdoc(s) under Other Personnel below.

Name of Student/Postdoc Investigator Degree

William Morrison

**Fmail** Phone

Fax

wmorrison@berkeley.edu

Department Name

Mailing Address


Protocol # 2020-08-13558 **PROTOCOL** Date Printed: 08/17/2021 Soc-Behav-Ed Exempt Berkeley Protocol Title: Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened beverages Soc-Behav-Ed Exempt Protocol Type: 06/27/2021 Date Submitted: This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details. Important Note: The Social Science Matrix UCB status (select all that apply): Faculty Postdoc X Grad Undergrad Other Faculty (with some exceptions), staff, and students engaged in human subjects research must complete either the biomedical or social-behavioral human research course through the online Collaborative Institutional Training Initiative (CITI), depending upon which is most germane to the research. ALL PIs on an NIH award are required to complete either CITI or NIH Training. See Training and Education for more information. If applicable, please insert date (mm/dd/yy) of completion in appropriate box(es) below: Other Training (title & date completed) CITI NIH 07/20/19


Protocol # 2020-08-13558 **PROTOCOL** Soc-Behav-Ed Exempt Berkeley Date Printed: 08/17/2021 Protocol Title: Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened beverages Protocol Type: Soc-Behav-Ed Exempt Date Submitted: 06/27/2021 This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details. Important Note: \* \* \* Vulnerable Subject Checklist \* \* \* Vulnerable Subject Checklist Yes No N Children/Minors N Prisoners Pregnant Women N N Fetuses N Neonates Educationally Disadvantaged N **Economically Disadvantaged** N N Cognitively Impaired Other (i.e., any vulnerable subject population(s) not specified above)


Protocol # 2020-08-13558 Date Printed: 08/17/2021

Protocol Title:

Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened

beverages

Protocol Type:

Soc-Behav-Ed Exempt

Date Submitted:

06/27/2021

Important Note:

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

\* \* \* Study Sites \* \* \*

#### Study Sites

Select all study sites where data collection via subject interaction will take place:

International

International Site(s) (specify country, region, and township or village)

Local

UC Berkeley

**UC Davis** 

**UC Irvine** 

UC Los Angeles

**UC Merced** 

UC Riverside

UC San Diego

UC San Francisco

UC Santa Barbara

UC Santa Cruz

Lawrence Berkeley National Laboratory

Alameda Unified School District (specify schools below)

Berkeley Unified School District (specify schools below)

Oakland Unified School District (specify schools below)

Other (Specify other Study Sites) X

The studies will take place online through the UC Berkeley-licensed version of Qualtrics.


**PROTOCOL** Soc-Behav-Ed Exempt Berkeley Protocol Title: Protocol Type: Date Submitted: Important Note:

Protocol # 2020-08-13558 Date Printed: 08/17/2021

Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened

beverages

Soc-Behav-Ed Exempt

06/27/2021

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

#### \* \* \* General Checklist \* \* \*

#### General Checklist

## Yes No

Is the research receiving any federal funding (e.g., NIH, NSF, DOD, etc.)?

Is another campus relying on UC Berkeley for IRB review by means of the UC System Memorandum of Understanding (MOU)?

Is another institution relying on UC Berkeley for IRB review by means of an Inter-institutional IRB Authorization Agreement?

Will subjects be compensated for participation?

Will any type of deception or incomplete disclosure be used? If yes, submit a non-exempt application.

Do investigators have a Conflict of Interest (COI)? If yes, submit a non-exempt application.


Protocol # 2020-08-13558 Date Printed: 08/17/2021

Protocol Title:

Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened

beverages

Protocol Type:

Soc-Behav-Ed Exempt

Date Submitted:

06/27/2021

Important Note:

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

\* \* \* Funding \* \* \*

#### **Funding Checklist**

NOTE: Only the Principal Investigator (PI) of the grant or subcontract can add his or her own SPO Funding information in this section. The PI of the grant must also be listed in the Personnel Information section of the protocol in one of the following roles: Principal Investigator or Faculty Sponsor, Student or Postdoctoral Investigator, Co-Principal Investigator, Administrative Contact, or Other Contact. Training Grants can be added by anyone in one of the aforementioned roles. For step-by-step instructions, see Add SPO Funding Quick Guide

Not Funded

SPO - Funding

## Funding - Other

| Funding<br>Type | Funding<br>Type | Sponsor/<br>Provider | # | Title | Amount | Begin | on | Lead PI<br><br><br>(If<br>different<br>from<br>Protocol<br>PI) |
|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|

## Funding - Other

**Funding Type** 

Other

PI Research Funds

Sponsor/Provider

Title Amount Begin End

Narrative Description

Dmitry Taubinsky's research funds. These will be used to fund the fuel economy survey.


PROTOCOL Soc-Behav-Ed Exempt Berkeley Protocol # 2020-08-13558 Date Printed: 08/17/2021 Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened beverages Protocol Title: Protocol Type: Soc-Behav-Ed Exempt Date Submitted: 06/27/2021 This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details. Important Note: Lead PI (If different from Protocol PI) Funding Type Other Funds from NBER Sponsor/Provider Title **Amount** Begin End We were awarded, through the NBER, an NIH grant to fund the sugar-sweetened beverages survey. The funds will remain at NBER who will directly compensate the participants. Narrative Description Lead PI (If different from Protocol PI)


Protocol # 2020-08-13558 Date Printed: 08/17/2021

Protocol Title:

Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened

beverages

Protocol Type: Soc-Behav-Ed Exempt

Date Submitted: 06/27/2021

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details. Important Note:

### \* \* \* Exempt Paragraph(s) \* \* \*

#### Exempt Paragraphs

Federal Policy for the Protection of Human Subjects (45 CFR 46) identifies categories of research activities involving human subjects that may be exempt from some of the requirements of subcommittee (expedited) or full committee review. In addition, UCB utilizes flexibility within the regulations to allow certain non-federally regulated activities to be exempted under UCB-defined category #70 (formerly #7). For more information and examples of exempt research, see <a href="https://cphs.berkeley.edu/exempt.pdf">https://cphs.berkeley.edu/exempt.pdf</a> target=blank > CPHS Guidelines on Exempt Research.

Exempt determinations must be made by OPHS Staff and the research must not begin until you have received notification that the research was determined to be exempt.

Select one or more of the following exempt categories. If research activities do not fit into one or more exempt categories, complete a non-exempt application.

NOTE: Certain research activities are not eligible for exempt status because additional protection has been required by federal regulations for vulnerable populations. Specifically, the following do not qualify for exempt status: (1) survey or interview of children; (2) observation of the public behavior of children when investigators interact with the children; (3) interactions with children; and (4) research involving prisoners except for research aimed at involving a broader subject population that only incidentally includes prisoners.

- EDUCATIONAL PRACTICES: Research, conducted in established or commonly accepted educational settings, that specifically involves normal educational practices that are not likely to adversely impact student's opportunity to learn required educational content or the assessment of educators who provide instruction. This includes most:
  - i) Research on regular and special education instructional strategies: OR
  - ii) Research on the effectiveness of or the comparison among instructional techniques, curricula, or classroom management methods.

\*This category does not apply to use of school records of identifiable students or interviewing instructors about specific students.

- EDUCATIONAL TESTS (COGNITIVE, DIAGNOSTIC, APTITUDE, ACHIEVEMENT), SURVEY PROCEDURES, INTERVIEW PROCEDURES, OR OBSERVATION OF PUBLIC BEHAVIOR (INCLUDING VISUAL OR AUDITORY RECORDING): Research involving these procedures is 2. exempt, IF one of the following is correct:
  - I) Any information obtained is recorded in such a manner that subjects CANNOT be identified, directly or through identifiers linked to the subjects; OR


Protocol # 2020-08-13558 Date Printed: 08/17/2021

Protocol Title:

Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened

beverages

Protocol Type:

Soc-Behav-Ed Exempt

Date Submitted:

06/27/2021

Important Note:

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

ii) Any disclosure of the subject's responses outside of the research could NOT reasonably place the subject at risk of criminal or civil liability or be damaging to the subject's financial standing, employability, educational advancement, or reputation; OR

iii) Any information obtained is recorded by the investigator in such a manner that the identity of the human subjects CAN readily be identified, directly or through identifiers linked to the subjects, AND an IRB conducts a limited IRB review to make the determination required by 45 CFR 46.111(a)(7).

"Workplace meetings and activities, as well as classroom activities, are not considered "public behavior."

RESEARCH INVOLVING BENIGN BEHAVIORAL INTERVENTIONS in conjunction with the collection of information from adult subjects through verbal or written response (including data entry) or audiovisual recording, if the subject prospectively agrees to the intervention and information collection, is exempt, IF: X

i) Any information obtained is recorded by the investigator in such a manner that the identity of the human subjects cannot readily be identified, directly or through identifiers linked to the subjects;

- X ii) Any disclosure of the subject's responses outside of the research could NOT reasonably place the subject at risk of criminal or civil liability or be damaging to the subject's financial standing, employability, educational advancement, or reputation; OR
  - iii) Any information obtained is recorded by the investigator in such a manner that the identity of the human subjects CAN readily be identified, directly or through identifiers linked to the subjects, AND an IRB conducts a limited IRB review to make the determination required by 45 CFR 46.111(a)(7).
- Secondary research for which consent is not required: Secondary research uses of identifiable private information or identifiable biospecimens, if at least one of the following criteria is met:
  - i) The identifiable private information or identifiable biospecimens are publicly available; OR
  - ii) The information is recorded by the investigator in such a manner that subjects cannot be identified, directly or through identifiers linked to the subjects, and the investigator does not contact or re-identify subjects; OR
  - iii) Exempt category 4iii is not in use at UC Berkeley.


Protocol # 2020-08-13558 Date Printed: 08/17/2021

Protocol Title:

Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened

beverages

Protocol Type:

Soc-Behav-Ed Exempt

Date Submitted:

06/27/2021

Important Note:

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol.

Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

iv) The research is conducted by, or on behalf of, a Federal department or agency using government-generated or government-collected information obtained for nonresearch activities, if government-generated or government-collected information obtained for nonresearch activities, in the research generates identifiable private information that is or will be maintained on information technology that is subject to and in compliance with section 208(b) of the E-Government Act of 2002, 44 U.S.C. 3501 note, if all of the identifiable private information collected, used, or generated as part of the activity will be maintained in systems of records subject to the Privacy Act of 1974, 5 U.S.C. 552a, and, if applicable, the information used in the research was collected subject to the Paperwork Reduction Act of 1995, 44 U.S.C. 3501 \*et seq.\*

- Research and demonstration projects that are conducted or supported by a Federal department or agency, or otherwise subject to the approval of department or agency heads (or the approval of the heads of bureaus or other subordinate agencies that have been delegated authority to conduct the neads of bureaus or other subordinate agencies that have been delegated authority to conduct the research and demonstration projects), and that are designed to study, evaluate, improve, or otherwise examine public benefit or service programs, including procedures for obtaining benefits or services under those programs, possible changes in or alternatives to those programs or procedures, or possible changes in methods or levels of payment for benefits or services under those programs. Such projects include, but are not limited to, internal studies by Federal employees, and studies under contracts or consulting arrangements, cooperative agreements, or grants. Exempt projects also include waivers of otherwise mandatory requirements using authorities such as sections 1115 and 1115A of the Social Security Act, as amended.
  - i) Each Federal department or agency conducting or supporting the research and demonstration projects must establish, on a publicly accessible Federal Web site or in such other manner as the department or agency head may determine, a list of the research and demonstration projects that the Federal department or agency conducts or supports under this provision. The research or demonstration project must be published on this list prior to commencing the research involving human subjects.
- TASTE AND FOOD QUALITY EVALUATION AND CONSUMER ACCEPTANCE STUDIES: This research is exempt, IF:
  - i) Wholesome foods without additives are consumed; OR
  - ii) A food is consumed that contains a food ingredient at or below the level and for a use found to be safe by the Food and Drug Administration (FDA) or approved by the Environmental Protection Agency (EPA) or the Food Safety and Inspection Service (FSIS) of the US Department of Agriculture (USDA); OR
  - iii) A food is consumed that contains an agricultural chemical or environmental contaminant at or below the level found to be safe by the FDA or approved by the EPA or the FSIS of the USDA.
- RESEARCH THAT INVOLVES NO GREATER THAN MINIMAL RISK TO SUBJECTS, BUT DOES NOT CONFORM TO A SPECIFIC EXEMPT CATEGORY UNDER 45 CFR 46.104(d) (exempt categories 1 through 6).


Protocol # 2020-08-13558 **PROTOCOL** Soc-Behav-Ed Exempt Berkeley Date Printed: 08/17/2021 Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened beverages Protocol Title: Protocol Type: Soc-Behav-Ed Exempt Date Submitted: 06/27/2021 This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details. Important Note: Category 70 minimal-risk exempt research activities that may include (but are not limited to) non-physically invasive interventions or performance of tasks. See CPHS guidelines on Exempt Research and Quick Guide for Exempt Category #70 for more information including exclusions and examples. 

Protocol # 2020-08-13558 Date Printed: 08/17/2021

Protocol Title:

Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened

beverages

Protocol Type: Soc-Behav-Ed Exempt

Date Submitted: 06/27/2021

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details. Important Note:

\* \* \* Purpose, Study Procedures and Background \* \* \*

Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened beverages

Complete Sections 1 - 9. Specify N/A as appropriate. Do not leave any required sections blank.

- 1. Purpose of the study
- Provide a brief explanation of the proposed research, including specific study hypothesis, objectives, and rationale.

The purpose of the research project is to explore the degree to which consumers tend to over-consume sugar-sweetened beverages or neglect fuel costs when purchasing cars. We propose to study these questions by conducting two surveys with "non-financial policy interventions" ("NPIs"), where we will provide select information to subjects and measure how the information alters their incentivized consumption behavior.

While the adverse health outcomes linked to sugar-sweetened beverage consumption affect all Americans, the impacts of these adverse health outcomes often manifest in old age. Cardiovascular disease is both the leading cause of death and the second leading cause of disability for older adults (Yazdanyar, 2010). Type 2 diabetes among elderly adults is associated with higher mortality, reduced functional status, and increased risk of institutionalization (Brown et al. 2003). Likewise, elderly obesity has been linked to increased risk of heart failure, impaired physical functionality, arthritis, cancers, and hypertension (Boateng et al., 2017). Additionally, obesity among younger adults may accelerate the aging process (Salvestrini et al., 2019) and is linked to increased risk of dementia later in life (Whitmer et al., 2005).

To study fuel costs, we will conduct a survey asking consumers to make hypothetical purchasing decisions for cars with different fuel efficiencies. We will have four treatment arms showing subjects one of the following: (i) the dollar value difference in gas costs between pairs of cars based on national averages of gas prices and miles driven per year, (ii) the dollar value difference in gas costs between pairs of cars based on the participant's self-reported gas price and miles driven per year, (iii) the MPG of each car, or (iv) which car is certified as environmentally friendly by the Environmental Protection Agency (via a " SmartWay Vehicle" logo).

To study sugar-sweetened beverages, we will conduct a survey asking consumers to make incentivized purchasing decisions for sugar-sweetened beverages. We will have three treatment arms showing subjects one of the following: (i) the nutrition label for the beverages, (ii) a warning label with text stating that consuming sugar-sweetened beverages can have adverse health consequences, and (iii) graphic warning label that shows images associated with diabetes, obesity, and tooth decay. We will also ask consumers to answer a series of nutrition knowledge questions, so that we can measure how the change in consumption behavior from an NPI correlates with their (lack of) nutritional knowledge.

2. Background


Protocol # 2020-08-13558 Date Printed: 08/17/2021

Protocol Title:

Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened

beverages

Protocol Type:

Soc-Behav-Ed Exempt

Date Submitted:

06/27/2021

Important Note:

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

Give relevant background (e.g., summarize previous/current related studies) on condition, procedure, product, etc. under investigation, including citations (with attached bibliography) if applicable.

Our project is related to several existing literatures. First, there are several studies which seek to quantify the effects of specific NPIs on purchasing behavior and wellbeing. One example is Allcott and Kessler (2019), which uses a field experiment to study the impact of home energy social comparison reports on consumer wellbeing. We will contribute by creating a comprehensive theoretical framework to understand whether an NPI is normatively good or bad. Using our online surveys, we will outline how to measure the relevant empirical parameters in practical settings. Second, we relate to a public health literature studying the effects of graphic warning labels on consumption for sugar-sweetened beverages, including Donnely et al. (2018) and Grummon et al. (2019).

Several of our survey questions also come from the existing literature. The nutrition questions Part I of our sugar-sweetened beverage survey were all previously used in Allcott, Lockwood, and Taubinsky (2019). Additionally, the warning labels used in Part II of our sugar-sweetened beverage survey were previously used in Grummon et al. (2019)

Our sugar-sweetened beverages survey also relates to an experimental economics literature that uses online shopping experiments. Sending participants the products is common economics experiments designed to simulate online shopping, and has been used in a variety of studies by members of this research team. Allcott and Taubinsky (2015) asks participants whether they would prefer environmentally friendly lightbulbs to standard lightbulbs at different prices, and send lightbulbs to participants based on their responses. Both Taubinsky and Rees-Jones (2018) and Morrison and Taubinsky (2020) have participants answer questions about whether or not participants would be willing to buy common household products at certain prices, and based on their responses, ship some participants products.

#### 3. Collaborative Research

If any non-UCB institutions or individuals are engaged in the research, explain their human research roles and what human subjects training they have/PI has planned to provide.

Dr. Hunt Allcott (Microsoft Research) is a coauthor in this project. He has completed the CITI training.

Dr. Allcott is involved in the study design, and will be involved in both the data analysis and drafting of the research paper.

Microsoft Research (MSR) is the academic research arm of Microsoft. MSR researchers regularly partner with university researchers, and Taubinsky and Allcott have been working together for 10 years. A link to MSR's economics research website is here: https://www.microsoft.com/en-us/research/research-

MSR is not providing research funding to UCB or UCB investigators. There is no consulting or business services agreement, and this is not a consulting or business services project.

MSR will defer to UCB for IRB review.

The National Bureau of Economic Research (NBER) was involved in applying for the NIH grant. Specifically, the NBER applies for an annual NIH grant that covers several projects, one of which is our sugar-sweetened beverages survey. The NBER is not involved in designing the survey, data collection, or


Protocol # 2020-08-13558 Date Printed: 08/17/2021

Protocol Title: Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened

beverages

Protocol Type: Soc-Behav-Ed Exempt

Date Submitted: 06/27/2021

Important Note:

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

data analysis. They also have no involvement in the fuel economy survey.

If any non-UCB institutions or individuals are collaborating in the research, complete the table below and b) attach any relevant IRB approvals in the Attachments section.

#### Non-UCB institutions

| Institution Name | Individual<br>Contact/ Affiliate<br>of Institution | FWA # | Local IRB<br>Review? (Y or<br>N) | IRB Approval<br>Date | IRB Approval<br>Expiration Date |
|---|---|---|---|---|---|
| Microsoft<br>Research (MSR) | Hunt Allcott | | N | | |
| National Bureau<br>of Economic<br>Research | Kristen Kenny | FWA00003692 | N (they wish to cede authority to the Berkeley IRB). | | |

#### 4. Study Procedures

Describe in chronological order of events how the research will be conducted, providing information about Describe in cironological order of events now the research will be conducted, providing information about all study procedures and who will conduct each (e.g., how participants are identified, the consent process, interventions/interactions with subjects, data collection), including follow-up procedures. If any interviews, questionnaires, surveys, or focus groups will be conducted for the study, explain and attach one copy each of all study instruments (standard and/or non-standard) in the Attachments section. Please see eProtocol Attachments Check List for Exempt Applications for more information. Indicate frequency and duration of visits/sessions, as well as total time commitment for participants in the study and an estimated time frame for when the study will be completed. If the proposed research involves secondary use of data/specimens, identified the proposed research involves secondary use of data/specimens. describe how data/specimens will be acquired

We will conduct two surveys, the first on fuel costs for cars and the second, two-part survey on sugarsweetened beverages.

For the fuel costs survey, the study population will consist of members of the AmeriSpeak Panel who choose to take our online survey.

For the sugar-sweetened beverages survey, we will use Facebook ads to recruit nationally-representative sample of people who are shopping online for soda, and direct them to a two-stage Qualtrics survey on the UC Berkeley licensed version of Qualtrics. We plan to use Facebook ads to target a larger section of adults aged 65 or older so that they comprise 25% of our total sample.

Qualtrics will provide us with de-identified data that contains the responses to the questions on our survey, the time taken for the total survey, and the time taken for each question of the survey. For the sugarsweetened beverages survey, we will collect their name, email address, and shipping address, in order to send them the compensation and bonuses. Investigators will not have access to any private Facebook


Protocol # 2020-08-13558 Date Printed: 08/17/2021

Protocol Title: Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened

beverages

Protocol Type: Soc-Behav-Ed Exempt

Date Submitted: 06/27/2021

Important Note:

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

send them the compensation and bonuses. Investigators will not have access to any private Facebook groups or accounts when posting Facebook ads.

For the fuel cost survey, AmeriSpeak will first draw the sample of potential participants, during which each potential participant will be assigned the linkage ID. Potential respondents will be invited to take the survey by an email from AmeriSpeak Support (as is typical for the platform), which will include a link to our standard AmeriSpeak survey platform, Voxco. This allows them to see that this is a legitimate, familiar AmeriSpeak study. The AmeriSpeak webpage on which they land will indicate that the survey is hosted by a partner site, and when the respondent clicks "Continue", they will be transferred to the UC Berkeley licensed version of Qualtrics. The link will have the anonymized ID post-pended to the link, so that the link "passes" the linkage ID to Qualtrics. This allows our research team to capture the linkage ID alongside the survey data collected in Qualtrics. AmeriSpeak will provide a redirect link back to the AmeriSpeak platform that the PI team will program at the end of the Qualtrics survey. The same ID number will be post-pended to that link, so Qualtrics "passes back" the linkage ID number. That allows AmeriSpeak to know who completed the survey and provide their corresponding demographics. Our research team will receive a file with the linkage ID, demographics and statistical weights. Respondents will not need to provide any linkage ID information, just answer the survey/experiment questions. These linkage IDs no purpose other than linking the demographics to the survey responses (and only to our survey responses; i.e., AmeriSpeak assigns creates a new set of linkage ID for each survey), and can only be linked to linked to any personal identifiable information via a key that only AmeriSpeak employees will have.

Separate workers will be recruited for the fuel cost survey and the sugar-sweetened beverage survey. Only participants who completed Part I of the sugar-sweetened beverage survey will be recruited to complete Part II.

For the fuel cost survey, Amerispeak will provide us with linkage IDs in order to link responses basic demographic information provided to us by AmeriSpeak.

Below we provide a brief description of each survey, copies of which are attached.

- I. Fuel cost cars survey
- Participants will first be given a brief description of the study and asked to provide their consent online via a yes/no question (they must select "yes" to continue). The consent form conforms to Berkeley guidelines. In particular, the consent form will include (i) the identity and affiliation of our research team, (ii) a clear description of the study procedures (including that they will be randomly assigned to one of several possible treatment arms) and how data will be used, (iii) a statement that this is a research study and that participation is voluntary, (iv) contact information from a member of our research team and for UC Berkeley CPHS for questions about the research, (v) the CPHS protocol ID number, and (vi) a notice that the research team will obtain their AmeriSpeak demographic survey responses from AmeriSpeak and link those demographic survey responses to their fuel cost survey responses. those demographic survey responses to their fuel cost survey responses.
- Participants will then answer some introductory questions, including listing their county and state of residence in 2019, estimating how many miles they drove with their primary vehicle in 2019, and estimating of gas costs per gallon in 2019.
- Participants will then be asked to rate four cars on a scale of 1-10 for how much they would like having the car. They are then asked to say how much they would be willing to pay for the car, if the gas were free.
- Participants are then given instructions for the rest of the survey, including how they can earn a bonus


Protocol # 2020-08-13558 Date Printed: 08/17/2021

Protocol Title:

Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened

beverages

Protocol Type:

Soc-Behav-Ed Exempt

Date Submitted:

06/27/2021

Important Note:

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

payment. Specifically, participants will be shown two cars and asked a series of questions about whether they would prefer to buy car A for \$X or car B for \$2,000. For each purchase, we compute a net annual value as:

o the maximum they told us earlier that they would pay per year to lease the car if gas is free, o minus the yearly gas cost, which is calculated with the car's official miles-per-gallon rating as well as the amount the participant reported driving in 2019 and the average gas price reported paying in 2019, o minus the yearly lease payment we quote below.

This net annual value is then rescaled so that the minimum bonus a participant can possibly earn is \$2, and the maximum is \$10.

- · Participants will then be shown two cars and asked a series of questions about whether they would prefer to buy car A for \$X or car B for \$2,000. They will answer these questions for two sets of cars.
- Participants will be shown two more sets of cars with additional information displayed on the screen (the "treatment"). All information provided will be true and factual. They will randomly be shown one of the following: (i) nothing (the control group: (i) the dollar value difference in gas costs between pairs of cars based on national averages of gas prices and miles driven per year, (ii) the dollar value difference in gas costs between pairs of cars based on the participant's self-reported gas price and miles driven per year, (iii) the MPG of each car, or (iv) which car is certified as environmentally friendly by the Environmental Protection Agency (via a "SmartWay Vehicle" logo). They will again answer a series of questions about whether they would prefer to buy car A for \$X or car B for \$2000.
- Total participation time is approximately 10-20 minutes to answer all the survey questions. Participants will be paid \$5 plus a bonus payment of \$2-\$10 for completing this survey.
- A copy of the survey guestions is attached (attachment\_survey\_cars).

#### II. Sugar-sweetened beverages survey

- Participants will first be given a brief description of the study and asked to provide their consent online via a yes/no question (they must select "yes" to continue). The consent form conforms to Berkeley guidelines. Participants will first be given a brief description of the study and asked to provide their consent online. The consent form conforms to Berkeley guidelines. In particular, the consent form will include (i) the identity and affiliation of our research team, (ii) a clear description of the study procedures (including that they will be randomly assigned to one of several possible treatment arms) and how data will be used, (iii) a statement that this is a research study and that participation is voluntary, (iv) contact information from a member of our research team and for UC Berkeley CPHS for questions about the research, and (v) the CPHS protocol ID number. They will also be told that we will ask for their email address, name, and shipping address in order to send them their rewards.
- · Participants will also be asked to enter their email address, which is how we will inform them to complete Part II of the survey.
- · Participants will then answer questions on basic demographic information (such as age, education, and income), their preferences for sugar-sweetened beverages, and a series of nutritional knowledge questions. This concludes Part I of the survey.
- At the end of Part I, participants will be told Part II that we will send a follow-up survey in 2-3 days via


Protocol # 2020-08-13558 Date Printed: 08/17/2021

Protocol Title:

Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened

beverages

Protocol Type: Soc-Behav-Ed Exempt

Date Submitted: 06/27/2021

Important Note:

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

#### email.

· After 2-3 days, participants will receive the follow-up survey. Only those who completed Part I will be eligible to complete this survey

- Participants will first be asked to give their consent again.
- Participants will then select their favorite sugar-sweetened beverages from a list.
- Participants Participants will be told they are shopping for sugar-sweetened beverages and asked to enter their name and the address where they want the product shipped.
- Participants will then be shown a picture of one of these sugar-sweetened beverages and a similar sugar free beverage (e.g., Minute Maid Lemonade and LaCroix Lemon). They will then answer a series of questions about whether they would prefer to buy the sugar-sweetened beverage for \$X or the sugar-free beverage for \$Y. Participants will answer these questions for three pairs of beverages, and are told they have a 1/3 chance of actually receiving beverages per one of their decisions.
- · Participants will then be shown three more pairs of beverages with additional information displayed on the screen (the "treatment"). All information provided will be true and factual. They will randomly be shown one of the following: (i) nothing (the control group), (ii) the nutrition labels for each beverage, (iii) a graphic warning label, or (iv) a warning label with text outlining negative health consequences of drinking beverages with added sugar.
- Total participation time is approximately 10-20 minutes to complete both parts of the survey. All questions for both parts of the survey are attached (attachment\_survey\_ssb\_part1 and attachment survey ssb part2)
- Participants will be paid \$6 for completing this survey: \$2 for completing part I and \$4 for completing part
- Additionally, all participants will receive an additional \$7.00 budget. For these participants, we will
  randomly choose one of the purchase decisions, and they will receive their choice of beverage (either the
  sugar-sweetened beverage or the sugar-free beverage) and \$7.00 minus the price of the drink. For
  example, if on the randomly chosen question, participants say they prefer Minute Maid Lemonade for
  \$4.50 to LaCroix Lemon for \$3.00, then they will receive the Minute Maid Lemonade and an additional

The procedure above ensures participants are incentivized to answer the questions as though they were really shopping for beverages in an online store. Sending participants the products is common economics really snopping for beverages in an online store. Sending participants the products is common economics experiments designed to simulate online shopping, and has been used in a variety of studies by members of this research team. Allcott and Taubinsky (2015) asks participants whether they would prefer environmentally friendly lightbulbs to standard lightbulbs at different prices, and send lightbulbs to participants based on their responses. Both Taubinsky and Rees-Jones (2018) and Morrison and Taubinsky (2020) have participants answer questions about whether or not participants would be willing to buy common household products at certain prices, and based on their responses, ship some participants

· Within 2-3 weeks from the end of the survey, we will ship the selected beverages to the participants using the shipping information they provide us.


Protocol # 2020-08-13558 Date Printed: 08/17/2021

Protocol Title: Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened

beverages

Soc-Behav-Ed Exempt Protocol Type:

Date Submitted: 06/27/2021

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details. Important Note:

• We include the 2-3 day waiting period between Parts I and II to minimize bias in the Part II responses. Without the waiting period, participants might be more inclined to focus on the nutritional aspects of the beverage than they would in their regular purchasing decisions.

State if photographing, audio, or video recording will occur and for what purpose (e.g. transcription, coding facial expressions). b)

Alternatives to Participation c)

Describe appropriate alternative resources, procedures, courses of treatment, if any, that are available to prospective subjects. If there are no appropriate alternatives to study participation, this should be stated. If the study does not involve treatment/intervention, enter "N/A" here.

NA

- If the proposed research involves secondary use of data/specimens, check all that apply: d)
  - i) coded private information or specimens, and the investigator will not have access to the key.
  - ii) from publicly available sources.
  - iii) recorded by the investigator in such a manner that subjects cannot be identified OR any link to identifying information has been destroyed.


Protocol # 2020-08-13558 Date Printed: 08/17/2021

Protocol Title:

Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened

beverages

Protocol Type:

Soc-Behav-Ed Exempt

Date Submitted:

06/27/2021

Important Note:

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

\* \* \* Subject Population \* \* \*

#### 5. Subject Population

Describe proposed subject population, including criteria for study inclusion and exclusion (e.g., age, health status, language, gender, race, ethnicity). State the maximum number of subjects planned for the study. This number should account for all subjects to be recruited, including those who may drop out or be found

For the sugar-sweetened beverages survey, our study population consists of participants recruited via Facebook ads who are shopping for soda. We aim to recruit a sample that will be broadly representative of the U.S. population in terms of race, gender, and education. We plan to overrecruit adults aged 65 or older so that they comprise approximately 25% of our sample. All U.S. residents aged 18 years or older will be eligible to enroll in our experiment.

For the fuel cost survey, our study population consists of AmeriSpeak panelists who own or are leasing a car. The survey will be advertised to AmeriSSeak panelists using a generic title (to avoid biasing respondents), as is common on these surveys: "Answer a 10-20 minute decision choice survey. You must own or be leasing a car to take this survey." All panelists are at least 18 years old. In addition, AmeriSpeak will work to ensure our subject population is nationally-representative along key demographics (race, gender, age, income, and education).

The maximum number of subjects planned for the study is 2,000 workers for the fuel cost survey and 3,000 workers for the sugar-sweetened beverages survey.


Protocol # 2020-08-13558 Date Printed: 08/17/2021

Protocol Title: Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened

beverages

Protocol Type: Soc-Behav-Ed Exempt

Date Submitted: 06/27/2021

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details. Important Note:

\* \* \* Risks \* \* \*

#### 6. Risks and Discomforts

Describe all known risks and discomforts associated with study procedures, whether physical, psychological, economic, or social (e.g., pain, stress, invasion of privacy, breach of confidentiality), noting probability and magnitude of potential harm.

The risk is an unintended breach of confidentiality, including due to possible third-party intervention online. We include a reminder to subjects at the end of the survey, i.e., the CPHS-recommended language: "You can help protect your privacy by clearing your browser's history, cache, cookies, and other browsing data. (Warning: This will also log you out of online services)."

If conducting educational tests, survey procedures, interview procedures, or observation of public behavior, AND linking to subjects' identifying information, explain why inadvertent release of the data would not have detrimental consequences (i.e. place subjects at risk of civil or criminal liability, or cause damage to their financial standing, employability or reputation). b)

For the sugar-sweetened beverages surveys, we will collect email address for the sole purpose of sending individuals Part II of the survey. We will also collect name and address so that we can ship them the

None of the data we receive is sensitive or could pose risk to the respondent if disclosed. We will only ask for the following information:

- Basic demographic information (age, race, sex, education, and income). Prospective participants will have the option to answer "prefer not to respond" for any of these questions.
   Self-assessment of frequency of sugary drink consumption, and related questions.
- · Knowledge about nutrition.
- · Preferences for sugar-sweetened beverages.

For the fuel economy survey, a linkage IDs in order to link responses basic demographic information provided to us by AmeriSpeak. These are unattached to any personal information, and serve no purpose other than linking the demographics to the survey responses. AmeriSpeak will then provide us with a file containing basic demographic information for these respondents (age, race, sex, education, and income), which we will then link to the survey responses. AmeriSpeak had previously surveyed all participants to obtain demographics, so essentially we are just linking the responses of two surveys.

None of the data we receive is sensitive or could pose risk to the respondent if disclosed. We will only receive the basic demographic information, and only ask for following information:

- Basic demographic information (age, race, sex, education, state/county of residence, and income).
- Self-assessment of environmental preferences.
  Preferences for different types of cars.
- In case of international research, describe the expertise you have, or have access to, which prepares you c) to conduct research in this location and/or with this subject population, including specific qualifications (e.g.,


Protocol # 2020-08-13558 **PROTOCOL** Soc-Behav-Ed Exempt Berkeley Date Printed: 08/17/2021 Protocol Title: Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened beverages Protocol Type: Soc-Behav-Ed Exempt Date Submitted: 06/27/2021 This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details. Important Note: to conduct research in this location and/or with this subject population, including specific qualifications (e.g., relevant coursework, background, experience, and training). Also, explain your knowledge of local community attitudes and cultural norms, and cultural sensitivities necessary to carry out the research. See CPHS Guidelines on Research in an International Setting.


Protocol # 2020-08-13558 Date Printed: 08/17/2021

Protocol Title: Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened

beverages

Protocol Type: Soc-Behav-Ed Exempt

Date Submitted: 06/27/2021

This Print View may not reflect all comments and contingencies for approval. Please check Important Note:

the comments section of the online protocol.

Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

#### \* \* \* Procedures to Maintain Confidentiality \* \* \*

#### 7. Confidentiality

NOTE: See CPHS Data Security Policy and CPHS Data Security Matrix before completing this section.

Will data be collected anonymously (i.e., no identifying information from subjects will be collected/ recorded that can be linked to the study data)? If no, please list all identifiable and/or coded data elements to be collected. Data is not anonymous if there is a code linking it to personally identifiable information. Also, audio and video recordings are generally not considered anonymous unless distinguishing features can be a) successfully masked.

For both surveys, we will set the Qualtrics to not collect IP addresses.

For the fuel cost survey, AmeriSpeak will provide us with linkage IDs so that (i) we can link individual responses to the basic demographic information sent to us by AmeriSpeak, and (ii) we can inform AmeriSpeak the bonus compensation each participant should be awarded. The research team will not have access to any identifiable information, but AmeriSpeak employees are able to link these linkage IDs to the participant's AmeriSpeak account. This link is necessary in order to provide the bonus compensation to these participants.

No member of our research team will have access to the key that links AmeriSpeak linkage IDs to the participant's AmeriSpeak account. These linkage IDs no purpose other than linking the demographics to the survey responses (and only to our survey responses; i.e., AmeriSpeak assigns creates a new set of linkage ID for each survey), and can only be linked to linked to any personal identifiable information via a key that only AmeriSpeak employees will have. It is not possible to determine the identify of an individual based on a combination of the data in the demographic information file.

For the sugar-sweetened beverage survey, we will collect their name and address so that we can ship participants their awarded beverages. We will also collect their email addresses so that we can send them Part II of the survey.

Explain how data, audiotapes, videotapes and photographs, etc. will be secured (e.g., password-protected computer, encrypted files, locked cabinet)stored and who will have access to them. Indicate at what point (b) they will be transcribed and/or destroyed (if ever).

All data will be downloaded from Qualtrics within one week of the end of data collection and deleted from Qualtrics within two weeks of the completion of the study.

Between Part I and Part II of the sugar-sweetened beverage survey, we will temporarily store the participants' email addresses on the researchers' password-protected UC Berkeley SharePoint account. The file containing this information will be encrypted, and will be destroyed within one week after we finish collecting responses for Part II. After Part II, we will also temporarily store their names and shipping information here. We plan to ship the beverages within 2-3 weeks from the end of the survey, and all PII will be destroyed once the beverages have been shipped.

Similarly, while waiting for the basic demographic information from AmeriSpeak, we will temporarily store


Protocol # 2020-08-13558 Date Printed: 08/17/2021

Protocol Title:

Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened

beverages

Protocol Type:

Soc-Behav-Ed Exempt

Date Submitted:

06/27/2021

Important Note:

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

the AmeriSpeak linkage IDs on the researchers' password-protected UC Berkeley SharePoint account. The file containing the IDs will be encrypted, and will be destroyed within one week after we receive the basic demographic information for these IDs from AmeriSpeak.

De-identified data will be retained indefinitely for possible use in future research done by ourselves or others. Participants will be informed of this during the consent process.


Protocol # 2020-08-13558 Date Printed: 08/17/2021

Protocol Title: Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened

beverages

Protocol Type: Soc-Behav-Ed Exempt

06/27/2021 Date Submitted:

Important Note:

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

\* \* \* Attachments \* \* \*

#### 8. Attachments

Add appropriate attachments (e.g. survey instrument(s), interview guide(s), reference list, other IRB approvals, etc.) in this section. Attachments must be in PDF or Word format. Please see eProtocol Attachments Check List for Exempt Applications for more information.

CITI Certificate(s)

| Document Type | Document Name |
|---------------------|---------------------------|
| CITI Certificate(s) | attachment_citi_morrison |
| CITI Certificate(s) | attachment_citi_taubinsky |

Inter-institutional Agreement

| Document Type | Document Name |
|-------------------------------|--------------------|
| Inter-institutional Agreement | MSR reliance form |
| Inter-institutional Agreement | NBER reliance form |

Questionnaire(s)

| Document Type | Document Name |
|------------------|------------------------------------|
| Questionnaire(s) | attachment amerispeak demographics |

## References

| Document Type | Document Name |
|---------------|-------------------------|
| References | attachment_bibliography |

Survey Instruments

| Document Type | Document Name |
|--------------------|-----------------------------|
| Survey Instruments | attachment_survey_cars |
| Survey Instruments | attachment_survey_ssb_part2 |
| Survey Instruments | attachment_survey_ssb_part1 |

Document Type CITI Certificate(s) Document Name attachment\_citi\_morrison

Document Type CITI Certificate(s) Document Name attachment\_citi\_taubinsky


Protocol # 2020-08-13558 Date Printed: 08/17/2021

Protocol Title:

Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened

beverages

Protocol Type:

Soc-Behav-Ed Exempt

Date Submitted:

06/27/2021

Important Note:

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

Document Type

Inter-institutional Agreement

**Document Name** 

MSR reliance form

Document Type

Inter-institutional Agreement

NBER reliance form

**Document Name** 

Questionnaire(s)

Document Type **Document Name** 

attachment\_amerispeak\_demographics

Document Type

References

**Document Name** 

attachment\_bibliography

Document Type Document Name Survey Instruments attachment\_survey\_cars

Document Type

Survey Instruments

**Document Name** 

attachment\_survey\_ssb\_part2

Document Type

Survey Instruments

Document Name

attachment\_survey\_ssb\_part1


Protocol # 2020-08-13558 Date Printed: 08/17/2021

Protocol Title: Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened

beverages

Protocol Type: Soc-Behav-Ed Exempt

Date Submitted: 06/27/2021

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details. Important Note:

\* \* \* Assurance \* \* \*

#### Assurance

As Faculty Sponsor, I understand that I am responsible for overseeing the protection of the rights and welfare of the human subjects, and adherence to CPHS requirements, federal regulations, and state statutes for this human subjects research.

#### I hereby assure the following:

- 1. I have read the protocol.
- 2. I have discussed with the Student/Postdoc Investigator how to comply with his or her assurances.
- 3. I will be available throughout the course of the study to provide guidance and consultation.
- I have read and agree to the above assurances.

As Student/Postdoctoral Investigator, I am responsible for the performance of this study, the protection of the rights and welfare of the human subjects, and strict adherence by all co-investigators and research personnel to CPHS requirements, federal regulations, and state statutes for this human subjects research.

## I hereby assure the following:

- The information provided in this application is accurate to the best of my knowledge.
- All experiments and procedures involving human subjects will be performed under my supervision or that of another qualified professional listed on this profocol.
- This protocol covers the human subjects research activities described in the grant proposal(s) (if applicable) supporting this research and any such activities that are not covered have been/will be covered by a CPHS approved protocol. 3.
- No change in the design, conduct, funding, or personnel of this research will be implemented without prior CPHS/OPHS review and approval.


Protocol # 2020-08-13558 Date Printed: 08/17/2021

Protocol Title: Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened

beverages

Protocol Type: Soc-Behav-Ed Exempt

06/27/2021 Date Submitted:

Important Note:

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

Participants' complaints or requests for information about the study will be addressed appropriately.

I will follow all relevant University of California system and UC Berkeley policies.

Should there be any changes that render this study <a class='PH1' href='javascript:getResearchExclusions()'>no longer eligible for exempt review, I will submit a new non-exempt application for CPHS review and approval. 7.

I have read and agree to the above assurances.


Protocol # 2020-08-13558 Date Printed: 08/17/2021

Protocol Title:

Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened beverages

Protocol Type: Soc-Behav-Ed Exempt

Date Submitted: 06/27/2021

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details. Important Note:

## \* \* \* Event History \* \* \*

## **Event History**

| Date | Status | View Attachments | Letters |
|---|---|---|---|
| 08/17/2021 | AMENDMENT 2 FORM APPROVED | Υ | Υ |
| 08/16/2021 | AMENDMENT 2 FORM SUBMITTED (CYCLE 3) | Υ | |
| 08/13/2021 | AMENDMENT 2 FORM<br>SUBMITTED (CYCLE 2) | Υ | |
| 07/16/2021 | AMENDMENT 2 FORM<br>SUBMITTED (CYCLE 1) | Υ | |
| 07/07/2021 | AMENDMENT 2 FORM<br>PANEL MANAGER<br>REVIEW | | |
| 06/27/2021 | AMENDMENT 2 FORM SUBMITTED | Υ | |
| 03/08/2021 | AMENDMENT 2 FORM CREATED | | |
| 02/03/2021 | AMENDMENT 1 FORM<br>APPROVED | Υ | Υ |
| 02/03/2021 | AMENDMENT 1 FORM SUBMITTED (CYCLE 3) | Υ | |
| 02/01/2021 | AMENDMENT 1 FORM SUBMITTED (CYCLE 2) | Υ | |
| 01/26/2021 | AMENDMENT 1 FORM SUBMITTED (CYCLE 1) | Υ | |
| 01/25/2021 | AMENDMENT 1 FORM<br>PANEL MANAGER<br>REVIEW | | |
| 01/22/2021 | AMENDMENT 1 FORM SUBMITTED | Υ | |
| 01/22/2021 | AMENDMENT 1 FORM CREATED | | |
| 09/14/2020 | NEW FORM APPROVED | Y | Υ |
| 09/10/2020 | NEW FORM<br>SUBMITTED (CYCLE 2) | Υ | |
| 09/04/2020 | NEW FORM<br>SUBMITTED (CYCLE 1) | Y | |


Protocol # 2020-08-13558 Date Printed: 08/17/2021

Protocol Title:

Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened beverages

Protocol Type:

Soc-Behav-Ed Exempt

Date Submitted:

06/27/2021

Important Note:

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

NEW FORM PANEL MANAGER REVIEW 09/01/2020

NEW FORM PANEL ASSIGNED 08/20/2020

**NEW FORM** 08/19/2020

SUBMITTED

08/17/2020 NEW FORM CREATED


Protocol # 2020-08-13558 Date Printed: 08/17/2021

Protocol Title:

Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened beverages

Protocol Type:

Soc-Behav-Ed Exempt

Date Submitted:

06/27/2021

Important Note:

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

Disclaimer: The generated PDF may not duplicate the original format completely. We do not warrant the accuracy of the changed format.

#### \* \* \* Attached Document \* \* \*

| Document Name | Created Date |
|------------------------------|--------------|
| attachment citi morrison.pdf | 03/08/2021 |




Protocol # 2020-08-13558 Date Printed: 08/17/2021

Protocol Title:

Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened beverages

Protocol Type:

Soc-Behav-Ed Exempt

Date Submitted:

06/27/2021

Important Note:

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

## \* \* \* Attached Document \* \* \*

| Document Name | Created Date |
|-------------------------------|--------------|
| attachment citi taubinsky.pdf | 03/08/2021 |






Completion Date 29-Dec-2017
Expiration Date N/A
Record ID 25627236

This is to certify that:

## **Dmitry Taubinsky**

Has completed the following CITI Program course:

Human Research (Curriculum Group)
Group 2 Social and Behavioral Research Investigators (Course Learner Group)
1 - Basic Course (Stage)

Under requirements set by:

University of California, Berkeley



Verify at www.citiprogram.org/verify/?wecedea79-c7e1-49b6-8582-771c36533ef3-25627236

Protocol # 2020-08-13558 Date Printed: 08/17/2021

Protocol Title:

Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened beverages

Soc-Behav-Ed Exempt Protocol Type:

06/27/2021 Date Submitted:

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details. Important Note:

## \* \* \* Attached Document \* \* \*

| Document Name | Created Date |
|-----------------------|--------------|
| MSR reliance form.pdf | 08/12/2021 |


## Committee for Protection of Human Subjects University of California, Berkeley

## REQUEST TO REVIEW RESEARCH FOR ANOTHER INSTITUTION

Non-UC reliances ONLY. To review for another UC IRB, see <u>UCB Reliance Registry</u>.

| Requirements<br>For UCB to revie | w for ano | her institution, ple | ase a | ffirm that the follo | owing is tr | rue: | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | do NOT have a p | | | | | ted with the | research. | |
| Relying Instituti | on | | | | | | | | |
| Institution Name | | Microsoft Resea | rch (N | MSR) | | | | | |
| This institution holds an active Federalwide Assurance (FWA). See FWA Lookup. FWA#: Click or tap here to enter text. | | | | | | ⊠ N/A | | | |
| Project | | | | | | | | | |
| Project Title: | Optimal | non-financial poli | cv inst | truments: fuel-eff | ficient car | s and sugar- | sweetened b | everages | |
| Reviewing IRB | Protocol N | Number: 2 | 020-0 | 8-13558 | | | | - | |
| | Funding<br>rt or attac | Source<br>h additional) | | UCB Re | UCB Recipient Status | | | SPO Award# | |
| Pl research fund | ds | | | ☐ Prime | □ Sub | ⊠ None | Click or tap here to enter tex | | |
| Funds from NBI | ER | | | ☐ Prime | □Sub | | Click or tap here to enter text | | |
| Click or tap here | e to enter | text. | | ☐ Prime | □ Sub | □ None | Click or tap here to enter tex | | |
| Click or tap here | Click or tap here to enter text. | | | | | □ None | Click or tap here to enter text. | | |
| | | nt of a federal awa<br>nts of another inst | | | subjects a | activities will | be carried | □ Yes | ⊠ No |
| UCB Investigate | ors | | | | | | | | |
| Principal Investi | igator: | | | Dmitry Taubinsky | | | | | |
| Co-/Student Investigator (if applicable): William Morrison | | | | | | | | | |
| Relying Investig | ators | | | | | | | | |
| Principal Investigator (must be eligible to | | | t Allcott | Email: | allcott@gmail.com | | | | |
| Co-/Student Investigator (if applicable): Click | | | | c or tap here to e | r tap here to enter text. Email: Click or tap here to e | | | here to ent | er text. |
| consent, adminis Dr. Hunt Allcott | tering inte | tive roles of collab<br>erventions, or anal<br>or in this project. He<br>ne research paper | yzing<br>le is ir | identifiable data) | , includin | g where they | will take pla | ice: | |
| The UCB Princip | al Investig<br>and <u>UCB</u> | elpal Investigator<br>pator agrees to co<br>Guidance on Relia | mply v | | | | | | 3 |
| Principal Invest | igator's S | Signature | | | | | Date | | |
| Version: 2/25/21 | | Please | subm | nit this form to op | hs@berke | eley.edu. | | F | Page <b>1</b> of <b>1</b> |

Version 1.0 – August 2021 Page **60** of **79** 

Protocol # 2020-08-13558 Date Printed: 08/17/2021

Protocol Title:

Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened beverages

Soc-Behav-Ed Exempt Protocol Type:

06/27/2021 Date Submitted:

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details. Important Note:

## \* \* \* Attached Document \* \* \*

| Document Name | Created Date |
|------------------------|--------------|
| NBER reliance form.pdf | 08/12/2021 |


## Committee for Protection of Human Subjects University of California, Berkeley

## REQUEST TO REVIEW RESEARCH FOR ANOTHER INSTITUTION Non-UC reliances ONLY. To review for another UC IRB, see <u>UCB Reliance Registry</u>.

| Requirements | for anot | har institution als | 2000 04 | firm that the fall | owing is to | | | | |
|---|---|---|---|---|---|---|---|---|---|
| For UCB to review | | ner institution, pie<br>do NOT have a r | | | | | ated with the | recearch | |
| □ NOTEOCD (es | ear of left | out NOT Have a p | Jolerili | ai iiilaiiolai <u>con</u> | mot of frite | assucia | ated with the | ieseaitii. | |
| Relying Institutio | n | | | | | | | | |
| Institution Name: | | National Bureau | of Eco | onomic Researd | ch | | | | |
| This institution holds an active Federalwide Assur See FWA Lookup. | | | | rance (FWA). | FWA#: | FWA00003692 | | | □ N/A |
| Project | | | | | | | | | |
| | Optimal | non-financial poli | cy inst | ruments: fuel-et | ficient cars | s and sugar | -sweetened b | peverages | |
| Reviewing IRB P | rotocol N | lumber: 2 | 020-08 | 8-13558 | | | | | |
| | unding :<br>or attac | Source<br>h additional) | | UCB Recipient Status | | | SPO Award# | | |
| PI research funds | 3 | | | ☐ Prime | □ Sub | | Click or tap here to enter te | | |
| Funds from NBEI | ₹ | | | ☐ Prime | □Sub | | Click or tap here to enter to | | |
| Click or tap here to enter text. | | | | ☐ Prime | □Sub | □ None | Click or tap here to enter to | | |
| Click or tap here | to enter | text. | | ☐ Prime | □Sub | □ None | Click or tap here to enter tex | | |
| | | nt of a federal awa | | | subjects a | activities will | be carried | □Yes | ⊠ No |
| out by employees | s or ager | its of another mst | itutiori | ŗ | | | | | |
| UCB Investigator | s | | | | | | | | |
| Principal Investig | mitry Taubinsky | / | | | | | | | |
| Co-/Student Inve | stigator | (if applicable): | V | Villiam Morrison | | | | | |
| Relying Investiga | tors | | | | | | | | |
| Principal Investigator (must be eligible to | | | en Kenny Email: | | | kennyk@nber.org | | | |
| Co-/Student Investigator (if applicable): Click | | | or tap here to | enter text. | . Email: | nail: Click or tap here to enter | | | |
| Roles Briefly describe the consent, administe | | | | | | | | | ng |
| The National Burapplies for an ani | eau of E<br>nual NIH<br>involved | conomic Researc<br>grant that covers<br>in designing the | h (NBE<br>sever | ER) was involve<br>al projects, one | d in applyi<br>of which i | ing for the N<br>s our sugar- | NIH grant. Spe-<br>sweetened b | ecifically, the | survey. |
| A | D Daine | in a l lacca ati a at a a | | | | | | | |
| Agreement by UC<br>The UCB Principal | | | | vith all requirem | ents and e | expectations | described in | UCB's IRE | 3 |
| Reliance Policy an | | | | | | | | | - |
| Dmitry Tau | binsk | y . | | | | | | | |
| 0 0 | | | | | | | August 12, | 2021 | |
| Principal Investig | ator's S | - | | SAN TANAN | | | Date | 100 | |
| Version: 2/25/21 | | Please | subm | it this form to or | ohs@berke | eley.edu. | | F | Page 1 of |

Version 1.0 – August 2021 Page **62** of **79** 

PROTOCOL Soc-Behav-Ed Exempt Protocol # 2020-08-13558 Date Printed: 08/17/2021 Berkeley Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened beverages Protocol Title: Protocol Type: Soc-Behav-Ed Exempt Date Submitted: 06/27/2021 This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details. Important Note: \* \* \* Attached Document \* \* \* Document Name Created Date attachment\_amerispeak\_demographics.pdf 03/08/2021

## **ATTACHMENT OMITTED - IRRELEVANT TO THIS PILOT**


Protocol # 2020-08-13558 Date Printed: 08/17/2021

Protocol Title:

Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened beverages

Protocol Type:

Soc-Behav-Ed Exempt

Date Submitted:

06/27/2021

Important Note:

This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details.

## \* \* \* Attached Document \* \* \*

| Document Name | Created Date |
|-----------------------------|--------------|
| attachment_bibliography.pdf | 08/12/2021 |


### References

- Allcott, H., Lockwood, B.B. & Taubinsky, D. (2019a). "Regressive Sin Taxes, with an Application to the Optimal Soda Tax," *Quarterly Journal of Economics* 134(3). DOI:10.1093/qje/qjz017
- Allcott, H., Lockwood, B.B & Taubinsky, D. (2019b). "Should We Tax Sugar-Sweetened Beverages? An Overview of Theory and Evidence," *Journal of Economic Perspectives* 33(3). DOI:10.1257/jep.33.3.202
- Allcott, H., & Kessler, J. (2019), "The Welfare Effects of Nudges: A Case Study of Energy Use Social Comparisons," *American Economic Journal: Applied Economics* 105(8)
- Donnelly, G.E., Zatz, L.Y, Svirsky, D. & John, L.K. (2018) "The Effect of Graphic Warnings on Sugary-Drink Purchasing," *Psychological Science* 29(8). PMID: 29912624
- Grummon, A. H., Hall, M. G., Taillie, L. S., & Brewer, N. T. (2019). "How Should Sugar-Sweetened Beverage Health Warnings be Designed? A Randomized Experiment." Preventive Medicine, 121. PMID: 30772370
- Grummon, A. H., Lockwood, B. B., Taubinsky, D., & Allcott, H. (2019). "Designing Better Sugary Drink Taxes." Science, 365(6457). PMID: 31488678
- Grummon, A. H., Taillie, L. S., Golden, S. D., Hall, M. G., Ranney, L. M., & Brewer, N. T. (2019). "Sugar-Sweetened Beverage Health Warnings and Purchases: A Randomized Controlled Trial." American Journal of Preventive Medicine, 57(5). PMID: 31586510
- Morrison, W & Taubinsky, D. (Forthcoming), "Rules of Thumb and Attention Elasticities: Evidence from Under- and Overreaction to Taxes," *Review of Economics and Statistics*.
- Taubinsky, D. & Rees-Jones, A (2018), "Attention Variation and Welfare: Theory and Evidence from a Tax Salience Experiment," *Review of Economic Studies*. 85(1).

PROTOCOL Soc-Behav-Ed Exempt Protocol # 2020-08-13558 Date Printed: 08/17/2021 Berkeley Optimal non-financial policy instruments: fuel-efficient cars and sugar-sweetened beverages Protocol Title: Protocol Type: Soc-Behav-Ed Exempt 06/27/2021 Date Submitted: This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details. Important Note: \* \* \* Attached Document \* \* \* Document Name Created Date 03/08/2021 attachment\_survey\_cars.pdf

## ATTACHMENT OMITTED - IRRELEVANT TO THIS PILOT

